CLINICAL TRIAL: NCT01529138
Title: Phase I Study of Axitinib and Temsirolimus in Solid Tumors
Brief Title: Study of Axitinib and Temsirolimus in Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Emory University (Other)
Collaborators: Pfizer (Industry)
Responsible Party: Principal Investigator, Bradley Carthon MD, PhD, Principal Investigator, Emory University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IRB00048705; WCI1939-10 (Other: Other)
Record Dates: First submitted 2011-11-14; First posted 2012-02-08 (Estimated); Last update posted 2015-04-13 (Estimated); Status verified 2015-04

CONDITIONS: Cancer
Keywords: Cancer
MeSH Terms: conditions — Neoplasms | interventions — Axitinib; temsirolimus

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Temsirolimus (Experimental): An ester of the macrocyclic immunosuppressive agent sirolimus.
  Interventions: Drug: Temsirolimus
- Axitinib (Experimental): An oral, selective inhibitor of vascular endothelial growth factor (VEGF) receptors 1, 2, 3.
  Interventions: Drug: Axitinib

INTERVENTIONS:
Drug: Axitinib — Combination treatment with temsirolimus and axitinib
  Other Names: Inlyta; AG013736
  Arms: Axitinib
Drug: Temsirolimus — Combination treatment with temsirolimus and axitinib
  Other Names: Torisel; CCI-779
  Arms: Temsirolimus

SUMMARY:
This study is being done to determine the highest safe dose of the combination of temsirolimus and axitinib; to learn the side effects when these drugs are given together; and to determine how the patient's disease responds to treatment.

The combination of the drugs temsirolimus and axitinib has not been studied before so it is unknown whether this treatment will have any benefit in the patient's cancer.

Temsirolimus is commercially available and approved for treatment of some types of kidney cancer.

Axitinib has been tested in several diseases but it is not yet commercially available for the treatment of any cancer in the United States.

The combination of temsirolimus and axitinib is not approved for treatment of any cancer outside of a clinical trial.

ELIGIBILITY:
Inclusion Criteria/Exclusion Criteria:

* Patients must have histologically confirmed non-hematologic malignancy for which standard curative or palliative measures do not exist or are no longer effective
* Patients with hepatocellular carcinoma do not need histologic confirmation of malignancy if the following criteria were met at diagnosis:

  * Liver lesions 1 - 2 cm with arterial enhancement and washout in venous phase of CT/MRI
  * Liver lesions ≥ 2 cm with arterial enhancement and washout in venous phase of CT/MRI or serum alpha-feto protein ≥ 200 ng/mL
* Eastern Cooperative Oncology Group (ECOG) Performance Status 0 or 1
* Marrow and Organ function requirements:

  * Absolute Neutrophil Count ≥ 1000/mm³
  * Platelets ≥ 75,000/mm³
  * Hemoglobin ≥ 9.0 g/dL
  * Total bilirubin ≤ 1.5 x upper limit of normal (ULN)
  * Alkaline phosphatase ≤ 2.5 x ULN (≤ 5 x ULN if liver metastasis present)
  * Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) ≤ 2.5 x ULN (≤ 5 x ULN if liver metastasis present or patient has diagnosis of hepatocellular carcinoma or cholangiocarcinoma)
  * Creatinine ≤ 1.5 x ULN
  * Urinalysis ≤ 1+ protein on dipstick or Urine creatinine:protein ratio < 1.0 If urine protein >1 1+ or urine creatinine:protein ratio > 1, then 24 hour urine protein should be obtained and the level should be < 1000 mg for patient enrollment.
  * Fasting serum cholesterol ≤ 350 mg/dL
  * Triglycerides ≤1.5 x ULN
* Life expectancy ≥ 12 weeks
* At least 2 weeks since end of prior systemic treatment (4 weeks for bevacizumab containing regimens), radiotherapy, or surgical procedure with resolution of all treatment related toxicity
* No evidence of uncontrolled hypertension as evidenced by 2 readings of < 140/90 measured 1 hour apart. Preexisting hypertension controlled with medication is allowed
* No gastrointestinal disorders including active peptic ulcer disease (within 6 months); active bleeding unrelated to malignancy; or melena, hematemesis, or hematochezia in the past 3 months without endoscopically-proven resolution
* No cardiovascular history within 12 months including: myocardial infarction (MI), uncontrolled angina, coronary artery bypass graft (CABG), or symptomatic congestive heart failure (CHF)
* Women of child bearing potential must have negative pregnancy test
* Willingness and ability to comply with scheduled visits
* Able to ingest oral medications
* No concurrent use or anticipated need for potent cytochrome P450 3A4 (CYP3A4) inhibitors or CYP3A4 or cytochrome P450 1A2 (CYP1A2) inducers

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2011-10; Primary Completion 2014-03 (Actual); Study Completion 2014-03 (Actual)

PRIMARY OUTCOMES:
Changes in the largest diameter (unidimensional measurement) of the tumor lesions and the shortest diameter in the case of malignant lymph nodes are used in the Response Evaluation Criteria in Solid Tumors (RECIST) criteria for evaluation. | Approximately re-evaluated every 8 weeks
  Complete Response: Disappearance of all target lesions.Any pathological lymph nodes must have reduction in short axis to <10 mm.
  Partial Response (PR): At least a 30% decrease in the sum of the diameters of target lesions Progressive Disease (PD): At least a 20% increase in the sum of the diameters of target lesions.Note: the appearance of one or more new lesions is also considered progressions).
  Stable Disease: Neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for PD.

CONTACTS AND LOCATIONS:
Overall Officials: Bradley Carthon, MD, PhD, Principal Investigator — Emory University Winship Cancer Institute
Locations (1):
- Emory University Winship Cancer Institute, Atlanta, Georgia, United States